CLINICAL TRIAL: NCT03111758
Title: Flow Augmentation With Geko Device in Patients With Postthrombotic Syndrome a Prospective Randomised Cross-Over Trial
Brief Title: Flow Augmentation Study in Postthrombotic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reaching total sample size was not feasible within the anticipated time frame.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NL59864.068.16
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Postthrombotic Syndrome
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Geko Device (Active Comparator): Neuromuscular Stimulator
  Interventions: Device: Flow augmentation
- IPCS (Active Comparator): Intermittent Pneumotic Compression Stocking
  Interventions: Device: Flow augmentation

INTERVENTIONS:
Device: Flow augmentation — Augmenting venous flow following deep venous stenting in patients with Postthrombotic syndrome

SUMMARY:
Rationale:

Stent therapy has been proven to be an effective form of therapy in the treatment of chronic iliofemoral and iliocaval post-thrombotic obstruction. During the first post-intervention day intermittent pneumatic compression stockings (IPCS) are necessary to augment venous flow. This will inherently prevent early stent occlusion. Our aim is to investigate whether the Geko device is effective as IPCS regarding augmentation of flow in post-thrombotic patients during the first day after stenting.

Objective: The primary objective of this study is to identify whether the Geko system is effective in augmenting flow compared to IPCS in post-thrombotic limbs before after stenting.

Study design: Interventional pilot study with randomized cross-sectional design.

Study population: Patients with a post-thrombotic obstruction undergoing a percutaneous procedure (PTA, stenting).

Intervention (if applicable): Treatment with intermittent pneumatic compression stockings (IPCS) and Geko-device.

Main study parameters/endpoints: The main endpoint and parameter of this study is time-averaged maximum flow velocity (TAMFV), measured by duplex ultrasonography using its pulse wave Doppler function.

ELIGIBILITY:
Inclusion Criteria:

* Post-thrombotic obstruction that requires percutaneous intervention through stenting, minimally 18 years of age

Exclusion Criteria:

* Peripheral arterial disease, comorbidities leading to impaired muscle function of either lower limb, co-morbidities affecting the circulatory system, history of deep venous surgery in either lower limb or groin, allergies to the plasters, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Time Averaged Maximum Flow Velocity | Five times one minute measurement
  time-averaged maximum flow velocity (TAMFV), measured by duplex ultrasonography (DUS) using its pulse wave Doppler function

CONTACTS AND LOCATIONS:
Overall Officials: Cees Wittens, MD,PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Summers JA, Clinch J, Radhakrishnan M, Healy A, McMillan V, Morris E, Rua T, Ofuya M, Wang Y, Dimmock PW, Lewis C, Peacock JL, Keevil SF. The geko electro-stimulation device for venous thromboembolism prophylaxis: a NICE medical technology guidance. Appl Health Econ Health Policy. 2015 Apr;13(2):135-47. doi: 10.1007/s40258-014-0139-0. PMID 25403719
- [Result] Williams KJ, Moore HM, Davies AH. Haemodynamic changes with the use of neuromuscular electrical stimulation compared to intermittent pneumatic compression. Phlebology. 2015 Jun;30(5):365-72. doi: 10.1177/0268355514531255. Epub 2014 Apr 10. PMID 24722790